CLINICAL TRIAL: NCT04268407
Title: 2-day Prophylactic Antibiotic is Effective in Transoral Endoscopic Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yichia Chan, principal investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902024A3
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Thyroid Nodule
Keywords: transoral surgery
MeSH Terms: conditions — Thyroid Nodule | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: thyroid nodules, plan for transoral thyroidectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-day prophylactic antibiotics (Experimental): use prophylactic antibiotic for 2 days after transoral thyroidectomy
  Interventions: Drug: Amoxicillin Clavulanate
- 7-day prophylactic antibiotic (Other): use prophylactic antibiotic for 7 days after transoral thyroidectomy
  Interventions: Drug: Amoxicillin Clavulanate

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — compare the duration of antbiotic use: 2 day versus 7 day
  Other Names: Augmentin

SUMMARY:
In transoral thyroidectomy via vestibular approach (TOETVA), prophylactic antibiotic for 5~7 days is recommended for the clean-contaminated wound. In this study, the investigators design a 2-day versus 7-day antibiotic prophylaxis to compare the surgical result and infection rate.

DETAILED DESCRIPTION:
Remote-access thyroid surgery has gained popularity and has advanced significantly over the past two decades, given the patient desire to avoid cosmetically displeasing scarring. The mostly recently introduced remote thyroid surgery is the transoral endoscopic thyroid surgery via vestibular approach (TOETVA). Because of the several advantages comparing with other removeaccess thyroid surgery, making it nowadays growing in popularity since 2016. However, TOETVA carry some inherent risks, including mental nerve injury, tumor seeding and local recurrence, fibrosis-induced long-lasting pulling sensation below the lower jaws, and surgical site infection coming from the clean-contaminated environment of oral incision.

Comparing with clean wound via the traditional open surgery, TOETVA carry the potential risk of infection. Based on the author's recommendation, prophylactic antibiotic (augmentin) will be administered 30 minutes before incision at operative room, followed by 2-day course of intravenous antibiotic, then shift to 5-day course of oral antibiotic finally. Up to date, only few case complicating postoperative infection were reported with extremely low infection rate (<1%). Therefore, the investigators want to study the short-course (2 days) of antibiotic coverage is also effective to prevent surgical site infection. It was proved in the preliminary study, comprising 5 patients in each group (2-day course in the study group and 7-day course in the control group). Later, the investigators will recruit more patients (n=100) to confirm this study.

ELIGIBILITY:
Inclusion Criteria:

1. Suspicious or proved thyroid cancer with size smaller than 4cm
2. Symptomatic benign thyroid nodules less than 6cm in size
3. Thyroid cyst
4. Follicular neoplasm
5. Graves' disease

Exclusion Criteria:

1. Previous thyroid or parathyroid surgery
2. History of radiation at neck
3. Could not tolerate the general anesthesia.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
post-operative infection | within one month after operation
  incidence of post-operative infection

SECONDARY OUTCOMES:
post-op complication | within one month after operation
  intensity of pain, measured by VAS(visual analogue score)

OTHER OUTCOMES:
post-op complication | within one month after operation
  mental nerve injury, measured by patient description of chin numbness
post-op complication | within one month after operation
  skin thermal or penetrated injury, noted during operation
post-op complication | within one month after operation
  post-operative hypoparathyroidism, measured by post-operative serum intact PTH level
post-op complication | within one month after operation
  recurrent laryngeal nerve injury, measured by clinical symptom and proved by laryngoscope

CONTACTS AND LOCATIONS:
Overall Officials: Yichia Chan, doctor, Principal Investigator — Kaohsing Chang Gung memorial hospital
Locations (1):
- Yi-Chia Chan, Kaohsiung City, 鳥松區, Taiwan

IPD SHARING:
Plan to Share IPD: No
only for request

REFERENCES:
- [Background] Anuwong A, Ketwong K, Jitpratoom P, Sasanakietkul T, Duh QY. Safety and Outcomes of the Transoral Endoscopic Thyroidectomy Vestibular Approach. JAMA Surg. 2018 Jan 1;153(1):21-27. doi: 10.1001/jamasurg.2017.3366. PMID 28877292
- [Background] Fernandez-Ranvier G, Meknat A, Guevara DE, Inabnet WB 3rd. Transoral Endoscopic Thyroidectomy Vestibular Approach. JSLS. 2019 Oct-Dec;23(4):e2019.00036. doi: 10.4293/JSLS.2019.00036. PMID 31719772
- [Background] Wang C, Zhai H, Liu W, Li J, Yang J, Hu Y, Huang J, Yang W, Pan Y, Ding H. Thyroidectomy: a novel endoscopic oral vestibular approach. Surgery. 2014 Jan;155(1):33-8. doi: 10.1016/j.surg.2013.06.010. Epub 2013 Jul 24. PMID 23890962